CLINICAL TRIAL: NCT00377728
Title: A 14 Day, Randomised, Double Blinded, Placebo-controlled 2-way Crossover Trial of Repeat Doses of Intranasal GSK256066 and Placebo in an Environmental Exposition Unit (Vienna Challenge Chamber) in Subjects With Seasonal Allergic Rhinitis (SAR)
Brief Title: Trial With Rhinitic Patients Taking GSK256066 Versus Placebo In A Pollen Challenge Chamber
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IPR101987
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Rhinitis, Allergic, Seasonal; Seasonal Allergic Rhinitis
Keywords: Seasonal Allergic Rhinitis Inflammation Vienna CHallenge Chamber
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — 6-((3-((dimethylamino)carbonyl)phenyl)sulfonyl)-8-methyl-4-((3-methyloxyphenyl)amino)-3-quinolinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK256066

SUMMARY:
This study is in patients with seasonal allergic rhinitis(SAR)and will compare the effect versus placebo of repeat doses of intranasal GSK256066 using the Vienna Challenge Chamber. GSK256066 is a potent and highly selective phosphodiesterase-4 (PDE4) inhibitor, currently in development by GSK for the treatment of allergic rhinitis, asthma and COPD.

Subjects will be selected on the basis that they display a defined moderate response to the pre-determined dose used. Opportunity to assess the efficacy of compounds versus placebo at maximal and trough plasma concentrations.

This study aims to explore the actions of repeat doses of intranasal GSK256066 in patients with Seasonal Allergic Rhinitis in the Vienna Challenge Chamber compared to placebo.

12-lead ECG, vital signs and adverse event enquiries will be made throughout the study. Nasal examination, symptom scores (TNSS), nasal lavage, nasal scrape and allergen challenge assessments will also be performed at various time points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects defined as individuals who are free from clinically significant illness or disease as determined by their medical history
* Body mass index less than 29.0 kg/m² with weight range of 55.0kg (females 50kg) to 95.0kg inclusive.
* History of seasonal allergic rhinitis
* Exhibit a moderate response to 1500 grass pollen grains/m3 after 2h in the Vienna Challenge Chamber
* Positive skin prick test for grass pollen at or within the 12 months preceding the screening visit.
* Positive RAST for grass pollen at or within the 12 months preceding the screening visit.
* Current non-smokers who have not used any tobacco products in the 6 months preceding the screening visit with a pack history of less than 10 pack years.
* Baseline FEV1 80% predicted and a baseline FEV1(maximum recorded value)/FVC(maximum recorded value) 70% predicted
* No conditions or factors which would make the subject unlikely to be able to stay in the chamber for 6 hours.
* Capable of giving informed consent which includes compliance with the requirements and restrictions listed in the consent form
* Available to complete all study measurements.

Exclusion Criteria:

* Pregnant or nursing females
* Women of childbearing potential who are unwilling or unable to use an appropriate method of contraception as outlined from at least two weeks prior to the first dose of study medication; and to continue until the final pregnancy test has been performed
* On examination the subject is found to have any structural nasal abnormalities or nasal polyposis, a history of frequent nosebleeds, recent nasal surgery or recent or ongoing upper respiratory tract infection which in the Responsible Physician's opinion renders the subject unsuitable for participation in the study
* Any respiratory disease other than mild stable asthma that is controlled with occasional use of as-needed short-acting beta-agonists and associated with normal lung function.
* The subject is likely to be unable to abstain from salbutamol use for 8 hours before a challenge
* The subject has a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* The subject has participated in a study with a new molecular entity during the previous 4 months or in any clinical study in the previous 3 months
* The subject is concurrently participating in another clinical study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.
* The subject has a screening QTc value of >430msec (>450msec for females), PR interval outside the range 120 to 240msec or an ECG that is not suitable for QT measurements
* The subject has donated a unit of blood (450mL) within the previous 3 months or intends to donate within 3 months of completing the study.
* The subject is currently taking regular (or a course of) medication whether prescribed or not, including steroids, vitamins, and herbal remedies Paracetamol and occasional as needed use of short-acting beta agonists is permitted.
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease*, * subjects will require normal serum creatinine clearance values at screening and normal serum creatinine value between 0.8 and 1.5 mg/dl
* The subject regularly, or on average, drinks more than 4 units of alcohol per day
* The subject is at risk of non-compliance with the study procedures/restrictions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2006-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Weighted mean total nasal symptom score (TNSS) (sneeze, itch, rhinorrhoea and obstruction) 0-6h post-dose period spent in the Vienna Challenge Chamber on Day 8 or 14

SECONDARY OUTCOMES:
Weighted mean nasal, eye and global symptom score and weighted mean nasal airflow resistance and secretion weight over 0-6 hours and 22-26h post dose on Day 8 (period 2 only) or Day 14 (period 1 only). FEV1, ECGs, AEs, and lab safety parameters

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Vienna, Austria